CLINICAL TRIAL: NCT06631963
Title: Telehealth Group-based Emotional Awareness and Expression Therapy for Patients With Persistent Physical Symptoms: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Maroti (Other)
Responsible Party: Sponsor-Investigator, Daniel Maroti, PhD, principal investigator, Stockholm University
Organization: Stockholm University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOSMOS3-Grupp
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Somatic Symptom and Related Disorders; Somatic Symptom Disorder; Functional Somatic Disorder; Functional Somatic Syndrome
MeSH Terms: conditions — Medically Unexplained Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group EAET delivered through telehealth (Other): Group-based Emotional Awareness and Expression Therapy (EAET) delivered through telehealth is a form of psychotherapy that helps individuals recognize and express emotions that may be contributing to physical symptoms. It is conducted in a group setting, allowing participants to share their experiences and support each other. Through a virtual platform, patients engage in structured sessions led by a therapist, where they explore emotional connections to their symptoms, practice emotional expression, and develop healthier coping mechanisms. The telehealth format enables access to therapy from remote locations, enhancing convenience and flexibility while maintaining the benefits of group interaction.
  Interventions: Behavioral: Emotional Awareness and Expression Therapy

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy — Emotional Awareness and Expression Therapy (EAET) is a form of psychotherapy designed to help individuals identify, process, and express emotions that may be linked to physical symptoms or chronic pain. It emphasizes the role of unresolved emotional experiences, such as trauma or interpersonal conflicts, in contributing to physical distress. Through EAET, patients learn to connect their emotions to their physical symptoms, express those emotions in a healthier way, and ultimately reduce both emotional and physical suffering. This therapy has been shown to be effective in treating conditions such as chronic pain, irritable bowel syndrome, and fibromyalgia.

SUMMARY:
Delivering Emotional Awareness and Expression Therapy (EAET) through digital or telehealth platforms in a group format offers several key advantages. First, it significantly improves access to care, allowing individuals with persistent physical symptoms (PPS) to receive effective, emotion-focused therapy regardless of their geographic location. Telehealth can also benefit those who face mobility issues or have limited access to specialized care in rural or underserved areas.

Group-based telehealth EAET promotes social connection among participants, fostering a supportive environment where individuals can share experiences, which may enhance therapeutic outcomes. Additionally, the convenience of remote therapy can reduce barriers to participation, such as time constraints and travel costs, making it easier for patients to commit to treatment.

Finally, the digital format allows for flexible, scalable interventions that can be easily integrated into routine psychiatric care, potentially increasing treatment uptake for individuals who might otherwise avoid in-person therapy due to stigma or logistical challenges.

ELIGIBILITY:
Inclusion Criteria:

* The participant certifies that he or she has undergone a medical evaluation for their physical symptoms (see separate certificate).
* The participant rates either moderate distress from physical symptoms on the PHQ-15 form (over 10 points) or significant distress from a single physical symptom (at least 2 points for that symptom).
* The participant expresses interest in exploring whether emotional factors, such as stress, may contribute to their symptom profile.
* Any prescribed medications must have been stable for at least 1 month.

Exclusion Criteria:

* Participants suffer from ongoing substance abuse (alcohol or drugs) or are assessed to have severe mental health issues (psychotic disorders, moderate to high suicide risk, antisocial personality disorder, etc.).
* Participants are currently prescribed medications that are clearly addictive and sedative in nature (e.g., benzodiazepines).
* Participants are involved in other psychological treatments focused on physical symptoms. However, other psychological treatments are allowed as long as the supportive therapy does not occur more than once a month.
* Participants do not have sufficient proficiency in the Swedish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionaire-15 (PHQ-15) | Change from pre to post treatment (i.e pre-treatment ca. 1 week before treatment. Post-treatment ca 1 week after treatment ends at 12 weeks.)
  Somatic symptom severity during the "last week" was assessed with the PHQ-15. Items were rated 0 ("Not bothered at all"), 1 ("Bothered a little"), or 2 ("Bothered a lot"); total scores range from 0 to 30 for women and 0-27 for men.
Visual Analoge Scales | Change from pre to post treatment (i.e pre-treatment ca. 1 week before treatment. Post-treatment ca 1 week after treatment ends at 12 weeks.)
  Visual Analoge Scales suggested by the EURONET-SOMA network (Rief et al., 2017). Somatic symptom intensity was measured from 1 ("No symptom") to 10 ("Symptom as bad as you can imagine") and somatic symptom interference from 1 ("No interference") to 10 ("Maximum interference").

SECONDARY OUTCOMES:
Patient Health Questionaire-9 (PHQ-9) | Change from pre to post treatment (i.e pre-treatment ca. 1 week before treatment. Post-treatment ca 1 week after treatment ends at 12 weeks.)
  PHQ-9 consists of nine questions withs ratings 0-3 (0= "not at all", 3= "almost every day") on impact of depressive symptoms. Higher scores indicate worse symptom/functioning with a maximum score of 27.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Change from pre to post treatment (i.e pre-treatment ca. 1 week before treatment. Post-treatment ca 1 week after treatment ends at 12 weeks.)
  GAD-7 consists of seven questions with ratings 0-3 (0= "not at all", 3= "almost every day") on impact of anxiety symptoms. Higher scores indicate worse symptom/functioning functioning with a maximum score of 21.
Post traumatic symptom Check List-5 (PCL-5) | Change from pre to post treatment (i.e pre-treatment ca. 1 week before treatment. Post-treatment ca 1 week after treatment ends at 12 weeks.)
  PCL-5 consists of 20 questions with ratings 0-4 on impact of post traumatic symptoms. Higher scores indicate worse symptom/functioning with a maximum score of 80.

OTHER OUTCOMES:
Negative Effects Questionnaire (NEQ) | At post-treatment (after 12 weeks of treatment)
  Participants respond to a series of statements regarding potential negative effects they may have experienced during or after therapy, typically using a Likert scale (e.g., 1 = "Not at all," to 5 = "Extremely"). The total score is computed by summing the responses, where higher scores indicate a greater frequency or severity of negative effects.
8 visual analogue scales | Mediational measure: Each week once a week throughout treatment, i.e. 11 measurement points. Week 2-12.
  A - 2 questions) Somatic symptom intensity was measured from 1 ("No symptom") to 10 ("Symptom as bad as you can imagine") and somatic symptom interference from 1 ("No interference") to 10 ("Maximum interference").
  B - 2 questions). On a scale 1-10 (as above) what is the capacity of emotional processing.
  C - 2 questions) On a scale 1-10 what is the capacity for self-compassion. D - 2 questions) On a scale 1-10 how much of symptoms is attributed to medical causes.
The Credibility and Expectancy Questionnaire (CEQ) | At treatment session 3 (out of 12)
  The CEQ includes items rated on a Likert scale (e.g., 1 to 9), where patients indicate their level of agreement with statements regarding the credibility and expected outcomes of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm University, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Participants has not approved this.